CLINICAL TRIAL: NCT04862806
Title: Safety, Efficacy and a Simple Model to Predict Response of BNT162b2 mRNA
Brief Title: Safety, Efficacy of BNT162b2 mRNA Vaccine in CLL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Ziv Medical Center (Other); Hadassah Medical Organization (Other); Ben-Gurion University of the Negev (Other); Galilee Medical Center (Unknown); Kaplan Medical Center (Other); Meir Medical Center (Other); Soroka University Medical Center (Other); Rambam Health Care Campus (Other); Sheba Medical Center (Other Government); Rabin Medical Center (Other); Sourasky Medical Center (Unknown)
Responsible Party: Principal Investigator, tamar.tadmor, HEAD OF HEMATOLOGY, Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0214-20-BNZ
Record Dates: First submitted 2021-03-21; First posted 2021-04-28 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; BNT162b2 mRNA Covid-19 Vaccine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Intervention Model Description: All enrolled CLL patients have received 2 shots of BNT162b2 mRNA vaccine, and the investigators will check the efficacy and safety of this vaccine in the enrolled population- the intervention is the diagnostic test of COVID-19 serology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Israel CLL study group (Experimental): BNT162b2 mRNA vaccine
  Interventions: Diagnostic Test: COVID-19 serology

INTERVENTIONS:
Diagnostic Test: COVID-19 serology — Immune response to BNT162b2 mRNA vaccine is assessed on the basis of anti covid19 IgG levels. A centralized assessment of the serological response for 4 medical centers is performed on serum samples stored at -60 °C using Abbott-SARS-CoV-2 IgG quant (Positive value > 151; range 0-40.000). The other 4 medical centers performed the test locally using DiaSorins-LAISISON SARS-CoV S1/S2 IgG test (positive value >15 range 15-400). In the central virus laboratory at the Chaim Sheba Medical center the test was done by Elisa-RDB (positive value >1.1; range 1.1-10).

SUMMARY:
On behalf of the Israel CLL study group the investigators will evaluate the efficacy and safety of BNT162b2 mRNA Covid-19 Vaccine in patients with chronic lymphocytic leukemia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL was according to the IWCLL criteria
* All patients received two 30-μg doses of BNT162b2, administered intramuscularly 3 weeks apart. (Pfizer).

Exclusion Criteria:

* previous covid19 virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in the number of participants with BNT162b2 mRNA vaccine-related adverse events as assessed by a questionnaire relating to the development of patients' side effects to the vaccine, which was developed by study investigators. | 2-6 weeks after second vaccination, 3 months after second vaccination, 6 months after second vaccination
  Answers to the questionnaire are reported and described in a scale of 0-5, where zero indicates the lack of any side effect. Each patient is asked to complete the questionnaire on the same clinic visit when blood is drawn for serologic tests.
Antibody Persistence after Third Dose of BNT162b2 mRNA COVID-19 Vaccination in Serongative Patients with Chronic Lymphocytic Leukemia | 6 months
  To study the efficacy of booster vaccine in patients with CLL who are seronegative after first 2 vaccines

SECONDARY OUTCOMES:
Change in the immune response to BNT162b2 mRNA vaccine assessed on the basis of anti covid-19 IgG levels. | 2-6 weeks after second vaccination, 3 months after second vaccination, 6 months after second vaccination
  A centralized assessment of the serological response for 4 medical centers is performed on serum samples stored at -60 °C using Abbott-SARS-CoV-2 IgG quant (Positive value > 151; range 0-40.000). The other 4 medical centers performed the test locally using DiaSorins-LAISISON SARS-CoV S1/S2 IgG test (positive value >15 range 15-400). In the central virus laboratory at the Chaim Sheba Medical center the test was done by Elisa-RDB (positive value >1.1; range 1.1-10).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Hematology Division, Chaim Sheba Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herishanu Y, Rahav G, Levi S, Braester A, Itchaki G, Bairey O, Dally N, Shvidel L, Ziv-Baran T, Polliack A, Tadmor T, Benjamini O; Israeli CLL Study Group. Efficacy of a third BNT162b2 mRNA COVID-19 vaccine dose in patients with CLL who failed standard 2-dose vaccination. Blood. 2022 Feb 3;139(5):678-685. doi: 10.1182/blood.2021014085. PMID 34861036